CLINICAL TRIAL: NCT03271346
Title: Intensive Trauma Treatment for Children Exposed to Parental Conflict
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Trauma Institute & Child Trauma Institute (Other)
Collaborators: Gratis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-GRE-1
Record Dates: First submitted 2015-02-17; First posted 2017-09-05 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Conflict, Interparental; Trauma, Psychological
MeSH Terms: conditions — Psychological Trauma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: intensive trauma-focused therapy

SUMMARY:
The purpose of this study is to track outcomes of the investigator's therapy approach with children of separation/divorce who have been exposed to parental conflict.

ELIGIBILITY:
Inclusion Criteria:

* child between the ages of 6 - 16
* parent concerned re child's distress and behaviors related to custody, visitation, etc.
* parent has the legal authority to obtain treatment for the child
* parent and child fluent in English

Exclusion Criteria:

* as per clinical judgment of the PI during a telephone screening (interview of the referring parent), determination that the child is unlikely to be responsive to the intensive therapy format. This would typically be due to the child having a severe intellectual impairment, major dissociative disorder, etc.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children exposed to parental conflict and contested custody
Sampling Method: Non-Probability Sample
Enrollment: 4 (Estimated)
Dates: Start 2015-02; Primary Completion 2019-01-30 (Estimated); Study Completion 2019-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in CROPS following treatment | Pre-treatment, 2 weeks post-treatment, 2 months post-treatment
  Child (self-) Report of Posttraumatic Symptoms
Change in PROPS following treatment | Pre-treatment, 2 weeks post-treatment, 2 months post-treatment
  Parent Report of Posttraumatic Symptoms
Change in SUDS following treatment | Pre-treatment, 2 weeks post-treatment, 2 months post-treatment
  Subjective Units of Distress Scale
Change in PRS following treatment | Pre-treatment, 2 weeks post-treatment, 2 months post-treatment
  Problem Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Ricky Greenwald, PsyD, Principal Investigator — Trauma Institute & Child Trauma Institute
Locations (1):
- Trauma Institute & Child Trauma Institute, Northampton, Massachusetts, United States